CLINICAL TRIAL: NCT07220213
Title: FELLAShip to Better Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: The Worship Center Christian Church (Unknown)
Responsible Party: Principal Investigator, Nashira Brown, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300015137; UAB (Other Grant/Funding Number: UAB Center for Clinical and Translational Science and O'Neal Comprehensive Cancer Center)
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: High Blood Glucose; High Cholesterol; High Cholesterol/Hyperlipidemia; Blood Sugar; High; Obesity & Overweight; Diabetes Type 2
MeSH Terms: conditions — Hyperglycemia; Hypercholesterolemia; Hyperlipidemias; Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: randomized trial with intervention and control waitlist arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FELLAship (Experimental): FELLAship intervention participants will receive the 24-week intervention according to the curriculum, to be delivered by a health coach, personal trainer, and community health worker.
  Interventions: Behavioral: FELLAship
- Waitlist Control (No Intervention): Individuals in the waitlist control arm will not receive the intervention during the evaluation period. They will have access to the intervention post-evaluation period.

INTERVENTIONS:
Behavioral: FELLAship — TheFELLAship intervention, grounded in Social Cognitive Theory (SCT) and guided by the Socioecological Model (SEM), focuses on enhancing participants' skills, knowledge and beliefs, and self-efficacy to promote cardiovascular health (CVH). The program provides health education aligned with the Diabetes Prevention Program (DPP) and American Heart Association's Check. Change. Control. (AHA CCC) curriculum to support behavior change in diet, physical activity, tobacco use, sleep, and clinical care engagement. Team-based coaching and physical activity sessions strengthen behavioral confidence and skill application.
  Arms: FELLAship

SUMMARY:
The goal of this clinical trial is to evaluate the implementation and effectiveness of the FELLAship program-a church-based cardiovascular health (CVH) intervention-in Black men aged 35-70 who are at risk for heart disease, diabetes, obesity, and related conditions. The main questions this study aims to answer are:

* Does participation in the FELLAship program improve cardiovascular health metrics (e.g., blood pressure, cholesterol, blood sugar) and health behaviors among Black men at The Worship Center Christian Church (TWC)?
* What factors influence the adoption, delivery, and sustainability of the FELLAship program in a faith-based setting? Researchers will compare an immediate-start intervention group and a delayed-start (waitlist control) group to assess both short-term health outcomes and program implementation factors.

Participants will:

* Attend a 90-minute weekly session for 24 weeks, including 45 minutes of physical activity led by a certified trainer and 45 minutes of health education delivered by trained coaches.
* Receive one-on-one support from a community health worker to reduce barriers to care and engage with primary care.
* Complete biometric health screenings and surveys at baseline, 12 weeks, and 24 weeks to assess clinical and behavioral outcomes.
* Use a smartwatch, blood pressure cuff, and other tools to track progress in real time.
* Participate in exit focus groups or interviews to share feedback about the intervention.
* A subset of TWC leaders and interventionists (N=15) will also be interviewed to assess implementation, resource needs, and sustainability.

This study uses the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework to assess Reach, Effectiveness, Adoption, Implementation, and Maintenance, and aims to inform scalable strategies for improving CVH among Black men in trusted community settings.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Black men
* Age 18 or older
* LE8 (Life's Essential 8) score (threshold not specified, but implies "less than ideal" CVH)
* English speaking
* Resides in the Metropolitan Birmingham, Alabama area
* No physical activity restrictions imposed by a healthcare provider

Exclusion Criteria:

* Not identifying as Black and male
* Under age 18
* Non-English speakers
* Not living in the Birmingham, Alabama metro area
* Having a healthcare provider-imposed restriction on physical activity
* Ideal CVH (i.e., LE8 (Life's Essential 8) score above inclusion threshold)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 90 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Life's Essential 8 Overall Score | 24 Weeks
  Change from baseline in the Life's Essential 8 overall cardiovascular health score (range 0-100, higher scores indicate better cardiovascular health), assessed at 12 and 24 weeks.

SECONDARY OUTCOMES:
Change From Baseline in Life's Essential 8 Blood Pressure Score | 24 Weeks
  Change from baseline in the Life's Essential 8 blood pressure subscore (range 0-100, higher scores indicate better cardiovascular health), derived from systolic and diastolic blood pressure measured using an automated sphygmomanometer.
Change From Baseline in Life's Essential 8 Body Mass Index Score | 24 Weeks
  Change from baseline in the Life's Essential 8 body mass index subscore (range 0-100, higher scores indicate better cardiovascular health), calculated using measured height (inches) and weight (pounds) to derive BMI.
Change in Life's Essential 8 Diet (subjective) | 24 Weeks
  Change from baseline in the Life's Essential 8 diet subscore (range 0-100, higher scores indicate better cardiovascular health), measured using the 16-item Mediterranean Eating Pattern for Americans questionnaire.
Change From Baseline in Life's Essential 8 Blood Lipids Score | 24
  Change from baseline in the Life's Essential 8 blood lipids subscore (range 0-100, higher scores indicate better cardiovascular health), derived from non-HDL cholesterol measured from a blood sample.
Change From Baseline in Life's Essential 8 Blood Glucose Score | 24 Weeks
  Change from baseline in the Life's Essential 8 blood glucose subscore (range 0-100, higher scores indicate better cardiovascular health), derived from hemoglobin A1c measured from a blood sample.
Change From Baseline in Perceived Stress Score | 24 Weeks
  Change from baseline in perceived stress, measured using the Perceived Stress Scale (PSS) score.
Change in Life's Essential 8 Physical Activity (Self Reported) | 24 Weeks
  Change from baseline in the Life's Essential 8 physical activity subscore (range 0-100, higher scores indicate better cardiovascular health), derived from self-reported minutes of moderate or vigorous physical activity per week.
Change in Life's Essential 8 Physical Activity (Accelerometry) | 24 Weeks
  Change from baseline in the Life's Essential 8 physical activity subscore (range 0-100, higher scores indicate better cardiovascular health), derived from 7 days of accelerometry data collected using an ActiGraph device.
Change From Baseline in Life's Essential 8 Nicotine Exposure Score | 24 Weeks
  Change from baseline in the Life's Essential 8 nicotine exposure subscore (range 0-100, higher scores indicate better cardiovascular health), based on self-reported use of cigarettes or inhaled nicotine delivery systems.
Change From Baseline in Life's Essential 8 Sleep Health Score | 24 Weeks
  Change from baseline in the Life's Essential 8 sleep health subscore (range 0-100, higher scores indicate better cardiovascular health), measured using self-reported average hours of sleep per night.
Change From Baseline in Patient Activation Measure (PAM) Score | 24 Weeks
  Change from baseline in patient activation, measured using the Patient Activation Measure (PAM) score.
Change From Baseline in Health-Related Social Needs Score | 24 weeks
  Change from baseline in health-related social needs, measured using the Centers for Medicare and Medicaid Services Accountable Health Communities Health-Related Social Needs Screening Tool.
RE-AIM Adoption, Implementation, and Maintenance Indicators | 156 Weeks
  Adoption, implementation, and maintenance indicators of the FELLAship intervention, assessed using structured interviews, meeting documentation, and organizational records in alignment with the RE-AIM framework.

CONTACTS AND LOCATIONS:
Locations (1):
- The Worship Center Cristian Church, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a relatively small, community-based sample recruited from a single faith-based organization. Even with de-identification, there is a heightened risk that individuals could be re-identified based on demographic characteristics or other contextual details. To protect participant privacy and honor community trust, we will limit data access to the study team and approved partners under strict data security protocols.